CLINICAL TRIAL: NCT02249546
Title: Comparison of the Efficacy of Triple Therapy With or Without Acetylcysteine in the First Line of Helicobacter Pylori Infection- A Multicenter Randomized Comparative Trial
Brief Title: Efficacy of Acetylcysteine-containing Triple Therapy in the First Line of Helicobacter Pylori Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Professor, National Taiwan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201406074MINC
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetylcysteine + PPI-amoxicillin-clarithromycin (Experimental): N-acetylcysteine 600mg bid Dexlansoprazole 60mg qd Amoxicillin 1000mg bid Clarithromycin 500mg bid All for 14 days
  Interventions: Drug: N-acetylcysteine + PPI-amoxicillin-clarithromycin
- PPI-amoxicillin-clarithromycin (Active Comparator): Dexlansoprazole 60mg qd Amoxicillin 1000mg bid Clarithromycin 500mg bid All for 14 days
  Interventions: Drug: PPI-amoxicillin-clarithromycin

INTERVENTIONS:
Drug: N-acetylcysteine + PPI-amoxicillin-clarithromycin
  Arms: Acetylcysteine + PPI-amoxicillin-clarithromycin
Drug: PPI-amoxicillin-clarithromycin — Triple therapy
  Arms: PPI-amoxicillin-clarithromycin

SUMMARY:
Helicobacter pylori infection has been shown to be associated with the development of gastric cancer and peptic ulcer diseases. Eradication of H. pylori infection could reduce the occurence or recurrence of these diseases. The triple treatment including a proton pump inhibitor, clarithromycin, and amoxicillin or metronidazole to treat H pylori infection, proposed at the first Maastricht conference has become universal since all the consensus conferences and guidelines around the world recommended it. However, the eradication rate of clarithromycin-based triple therapy has been declining in recent years, probably related to the increasing resistant rate to clarithromycin. It was estimated that 15-20% of patients would fail from first line standard eradication therapy and need second line rescue therapy.

The H. pylori persistence in human infections and its resistance to the drugs commonly used in antimicrobial therapy have been attributed not only to genetic variability, but also to ability of H. pylori to form biofilm as a strategy to overcome environmental stress and to protect itself. Several recent reports indicate that H. pylori forms biofilm either in vitro or in vivo, N-acetylcysteine (NAC) were thought to reduce and prevent biofilm formation. Two small-scale clinical trials showed NAC offers additive effect on eradication effects of H. pylori therapy. A recent trial showed N-acetylcysteine pre-treatment before a culture-guided antibiotic regimen is effective in treating refractory H. pylori infection.

Aims: Therefore, we aim to assess

1. Whether triple therapy containing N-acetyl cysteine is more effective than standard triple therapy
2. the impact of antibiotic resistance and cytochrome P450 C19(CYP2C19) polymorphism on the eradication rate of triple therapy containing N-acetyl cysteine.

DETAILED DESCRIPTION:
Helicobacter pylori infection has been shown to be associated with the development of gastric cancer and peptic ulcer diseases. Eradication of H. pylori infection could reduce the occurrence or recurrence of these diseases. The triple treatment including a proton pump inhibitor, clarithromycin, and amoxicillin or metronidazole to treat H pylori infection, proposed at the first Maastricht conference has become universal since all the consensus conferences and guidelines around the world recommended it. However, the eradication rate of clarithromycin-based triple therapy has been declining in recent years, probably related to the increasing resistant rate to clarithromycin. It was estimated that 15-20% of patients would fail from first line standard eradication therapy and need second line rescue therapy. Measures to improved H. pylori eradication rate include (1) increase treatment duration, (2) add other antibiotics or use antibiotics not previously used, (3) introducing new therapeutic agents, and (4) potent acid inhibition. Our group has shown the 10- or 14-day sequential therapy, which consists of a proton-pump inhibitor and amoxicillin for the first 5 or 7 days, followed by a proton-pump inhibitor plus clarithromycin and metronidazole (or tinidazole) for another 5 or 7days, provides good eradication in first line H. pylori eradication. However, complexity of sequential therapy is complex and adverse effect resulted from adding one more antibiotic may have poor effect on compliance and leads to treatment failure. A simplified regimen for H. pylori infection is worthy of investigation.

Introducing new therapeutic agents The H. pylori persistence in human infections and its resistance to the drugs commonly used in antimicrobial therapy have been attributed not only to genetic variability, but also to ability of H. pylori to form biofilm as a strategy to overcome environmental stress and to protect itself. A biofilm is a dense aggregation of microbial cells bound together by a slimy extracellular matrix of polysaccharide and protein. When bacteria group together in these multicellular communities, they are able to tolerate antimicrobial challenges that normally eradicate free-floating individual cells. It is currently accepted that biofilms are implicated in over 80% of the chronic infections caused by bacteria, including middle ear otitis, endocarditis, urinary tract infections and lung infections of patients with cystic fibrosis. The importance of biofilm in medicine is due to its role in persistence of the infection because biofilm is not removed and bacteria in biofilms are 1000 more resistant to antibiotics and host defenses as compared to those free living bacteria.

Several recent reports indicate that H. pylori forms biofilm either in vitro or in vivo, Cole et al studied the ability of 19 H. pylori clinical isolates and reference strains in Brain Heart Infusion broth supplemented with 0.1% β-cyclodextrin. Both strains were able to form biofilm and the biofilm produced had a similar progression when compared to biofilm formed by other bacterial species. The first evidence of in vivo biofilm formation arose in 2006. The authors compared, by scanning electron microscopy, gastric biopsies from urease positive and negative patients, detecting the presence of dense mature biofilm in the pathogen positive biopsies while biofilm was absent in the urease negative biopsies, which is indicative that H. pylori is able to form biofilm in the human gastric mucosa. To this context, it is notable that stress conditions stimulate H. pylori to enter coccoid forms that when the antibiotic concentration reduces, can resuscitate and repopulate the biofilm and the infection relapses. In vitro study, H. pylori biofilm formation decreases the susceptibility to clarithromycin and that H. pylori clarithromycin resistance mutations are more frequently generated in biofilms than in planktonic cells.

Because antibacterial susceptibility of a particular strain is favored when the biofilm is destabilized, it is believed that a combination of antimicrobial agents and anti-biofilm molecules should be synergistic. N-acetylcysteine (NAC) being both a mucolytic agent and a thiol-containing antioxidant agent was successfully used in medical practice for the treatment of patients with chronic respiratory tract infections. The NAC positive effects were thought to be due not only to mucus-dissolving properties, but also, interestingly, to the capability to reduce and prevent biofilm formation. NAC was able to avoid biofilm formation and to destabilize the already formed biofilm at concentrations over 10 mg/mL, similar to results observed with other pathogens. On the other hand, in vivo studies with two groups of 20 individuals each, one group (treated) received N-acetyl-cysteine for one week before the anti-H. pylori treatment for refractory H. pylori infection while the other group (untreated controls) did not received the destabilizing agent, showed eradication of the infection in 65% of the cases for the N-acetyl-cysteine treated group as detected by the urea breath test. The control group showed only 20% of successful eradication, suggesting that N-acetyl-cysteine act as a biofilm destabilizing agent that favor in vivo the activity of antibiotic substances.

Potent acid inhibition Acid inhibition has also proven an important component of eradication therapy. The antibiotics, particularly clarithromycin, which is used against H. pylori, are subject to pH-dependent degradation. This degradation is reduced by increasing gastric pH. Achieving a pH above 4 maximizes the efficacy of the antibiotic. Second, proton pump inhibitors (PPIs) may alter the transport of antibiotics from the plasma to the gastric juice and mucosa by altering the pH or by affecting active transport processes. The minimum inhibitory concentration (MIC) of the antibiotics against H. pylori is often lower at higher pHs. Finally, because H. pylori is sensitive to changes in gastric pH, PPI-induced elevations of pH, the gastric contents may become less hospitable to H. pylori. The importance of achieving adequate acid inhibition has been highlighted by recent studies. First, increasing the PPI dose was found to raise cure rates when used in dual anti-Helicobacter pylori therapies. Second, a previous meta-analysis by our group showed that triple therapy using a standard dose of PPI twice a day achieves higher cure rates than the same antibiotics plus the PPI once daily. Previous meta-analyses show that H. pylori treatment achieves lower cure rates in extensive metabolizers than in poor PPI metabolizers. All this evidence supports the hypothesis that achieving a potent acid inhibition can improve cure rates of H. pylori treatment.

Lansoprazole, a proton pump inhibitor that specifically inhibits H+K+-ATPase in the gastric parietal cell, effectively inhibits both basal- and gastric-stimulated acid secretion. Our studies have proved lansoprazole-based H. pylori eradication achieved high successful rate. Dexlansoprazole modified release (MR), a new generation of proton pump inhibitor, is a novel modified release formulation of dexlansoprazole, an enantiomer of lansoprazole. Dexlansoprazole MR employs an innovative Dual Delayed Release (DDR) technology designed to prolong the plasma concentration-time profile of dexlansoprazole and extend the duration of acid suppression. In a phase 1 pharmacokinetic/pharmacodynamic study of Dexlansoprazole MR 60 and 90 mg once daily also produced significant increases in the percentage of time with intragastric pH >4 over 24-h postdose compared with lansoprazole 30 mg once daily (∼70% for dexlansoprazole MR vs. 60% for lansoprazole, P < 0.05). Since acid inhibition is crucial in H. pylori treatment. Whether a more potent PPI, Dexlansoprazole MR could improve the efficacy of H. pylori treatment has not been investigated.

Therefore, the primary purpose of the proposed study is to compare the efficacy of dexlansoprazole MR based triple therapy with or without N-acetyl cysteine for helicobacter pylori eradication

ELIGIBILITY:
Inclusion Criteria:

* H. pylori infected patients who have willingness to receive eradication therapy

Exclusion Criteria:

* (1) history of gastrectomy, (2)gastric malignancy, including adenocarcinoma and lymphoma, (3) previous allergic reaction to antibiotics (amoxicillin, clarithromycin), N-acetyl cysteine and prompt pump inhibitors (dexlansoprazole), (4)contraindication to treatment drugs, (5) pregnant or lactating women, (6) severe concurrent disease. (7) phenylketonuria (8) Patients who cannot give informed consent by himself or herself.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Helicobacter pylori eradication rate | 6wks

SECONDARY OUTCOMES:
Compliance | 14 days
Adverse effects | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, MD, PHD, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan Univeristy Hospital, Taipei, Taiwan
  - Department of Internal Medicine, National Taiwan Univeristy Hospital Yun-Lin branch, Douliu, Yunlin County

REFERENCES:
- [Derived] Chen CC, Luo JC, Fang YJ, Lee JY, Kuo CC, Yang TH, Chiu MC, Yu JJ, Bair MJ, Chen PY, Chou CK, Chen CY, Chang CY, Hsu YC, Tseng CH, Hsu WF, Hu WH, Tsai MH, Hsieh CL, Chen MJ, Shun CT, Liu TY, Lee YC, Liou JM, Wu MS; and for the Taiwan Gastrointestinal Disease and Helicobacter Consortium. Comparison of the effect of clarithromycin triple therapy with or without N-acetylcysteine in the eradication of Helicobacter pylori: a randomized controlled trial. Therap Adv Gastroenterol. 2020 Jul 31;13:1756284820927306. doi: 10.1177/1756284820927306. eCollection 2020. PMID 32821287